CLINICAL TRIAL: NCT03618368
Title: Second Clinical Evaluation of THERANOVA-500 Dialyzer in Chronic Hemodialysis (HD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Réseau de Santé Vitalité Health Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NEP2018-01
Record Dates: First submitted 2018-06-15; First posted 2018-08-07 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: End Stage Renal Disease on Dialysis

STUDY DESIGN:
Intervention Model Description: 1 blinded group on THERANOVA-500 dialyzer (Expanded Hemodialysis (HDx))
  1 blinded group on REVACLEAR-400 dialyzer (conventional hemodialysis (HD))
  1 non-blinded group on THERANOVA-500 dialyzer (Expanded Hemodialysis (HDx))
  1 non-blinded group on REVACLEAR-400 dialyzer (conventional hemodialysis (HD))
Who Masked: Participant
Masking Description: blinded group: as dialyzers are almost identical except for their labels, blinding is achieved by masking dialyzer labels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Blinded THERANOVA-500 dialyzer (Experimental): This group of 25 subjects is dialyzed with masked THERANOVA-500 dialyzer enabling Expanded Hemodialysis (HDx) therapy.
  Interventions: Device: THERANOVA-500 dialyzer
- Blinded REVACLEAR-400 dialyzer (Placebo Comparator): This group of 25 subjects is dialyzed with masked REVACLEAR-400 dialyzer enabling conventional hemodialysis (HD).
  Interventions: Device: REVACLEAR-400 dialyzer
- Unblinded THERANOVA-500 dialyzer (Experimental): This group of 10 subjects is dialyzed with unmasked THERANOVA-500 dialyzer which enables Expanded Hemodialysis (HDx) therapy.
  Interventions: Device: THERANOVA-500 dialyzer
- Unblinded REVACLEAR-400 dialyzer (Placebo Comparator): This group of 10 subjects is dialyzed with unmasked REVACLEAR-400 dialyzer which enables conventional hemodialysis (HD).
  Interventions: Device: REVACLEAR-400 dialyzer

INTERVENTIONS:
Device: THERANOVA-500 dialyzer — THERANOVA-500 dialyzer is a hemofilter that enables Expanded Hemodialysis (HDx) therapy.
  Arms: Blinded THERANOVA-500 dialyzer; Unblinded THERANOVA-500 dialyzer
Device: REVACLEAR-400 dialyzer — REVACLEAR-400 dialyzer is an usual hemofilter that enables conventional hemodialysis (HD).
  Arms: Blinded REVACLEAR-400 dialyzer; Unblinded REVACLEAR-400 dialyzer

SUMMARY:
Single blinded randomized controlled trial comparing Expanded Hemodialysis (HDx) using THERANOVA-500 dialyzer versus conventional hemodialysis (HD) using REVACLEAR-400 dialyzer in chronic hemodialysis patients over a 6-week intervention period. Primary endpoint is post-hemodialysis recovery time. Secondary endpoints are six pre-dialysis biomarker levels (b2-microglobuline, procalcitonine, free light chains (gamma-lambda), IL-6, CRP) and three Quality of Life (QoL)(adapted KDQoL-SF questionnaire, EQ-5D, and rESAS).

DETAILED DESCRIPTION:
This is a randomized controlled trial involving 70 subjects divided in 4 groups: 25 single blinded subjects using THERANOVA-500 dialyzer enabling Expanded Hemodialysis (HDx) ; 25 single blinded subjects using REVACLEAR-400 dialyzer enabling conventional hemodialysis (HD); 10 non-blinded subjects using THERANOVA-500 enabling Expanded Hemodialysis (HDx) and 10 non-blinded subjects using REVACLEAR-400 dialyzer enabling conventional hemodialysis (HD) for their chronic hemodialysis treatments over an active intervention period of 6 weeks. All subjects are to be dialyzed using REVACLEAR-400 enabling conventional hemodialysis (HD) for two weeks prior and for two weeks after the intervention period.

Primary endpoint is mean post-hemodialysis recovery time (as reported by subjects once weekly) between groups (THERANOVA-500 vs REVACLEAR-400) (all subjects) during the 6-week intervention period.

Secondary endpoints are:

1. Post-hemodialysis recovery time change (mean of 2-week pre and 2-week post intervention period compared to mean during 6-week intervention period)(mean THERANOVA-500 vs mean REVACLEAR-400)(all subjects),
2. Post-hemodialysis recovery time difference (mean between blinded and non-blinded THERANOVA-500 treated subjects during the 6-week intervention period,
3. Post-hemodialysis recovery time difference (mean between blinded and non-blinded REVACLEAR-400 treated subjects during the 6-week intervention period),
4. Post-hemodialysis recovery time difference mean gap between secondary endpoints 2 and 3,
5. Percentage of subjects who report no (zero) recovery time (mean THERANOVA-500 vs mean REVACLEAR-400) during 6-week intervention period (all subjects),
6. Pre and post 6-week intervention period pre-dialysis difference levels of beta-2 microglobulin (mean THERANOVA-500 vs mean REVACLEAR-400)(all subjects)(in nmol/L),
7. Pre and post 6-week intervention period pre-dialysis difference levels of procalcitonin (mean THERANOVA-500 vs mean REVACLEAR-400)(all subjects)(in ng/ml),
8. Pre and post 6-week intervention period pre-dialysis difference levels of free light chains (gamma and lambda)(mean THERANOVA-500 vs mean REVACLEAR-400)(all subjects)(in mg/L),
9. Pre and post 6-week intervention period pre-dialysis difference levels of interleukine-6 (mean THERANOVA-500 vs mean REVACLEAR-400)(all subjects)(in pg/ml),
10. Pre and post 6-week intervention period pre-dialysis difference levels of C reactive protein (CRP)(mean THERANOVA-500 vs mean REVACLEAR-400)(all subjects)(in mg/L),
11. Quality of life change (pre and at 2 weeks of intervention period) (mean THERANOVA-500 vs mean REVACLEAR-400)(all subjects)(assessed by adapted KDQoL-SF questionnaire)(max score 130),
12. Quality of life change (pre and at 4 weeks of intervention period) (mean THERANOVA-500 vs mean REVACLEAR-400)(all subjects) assessed by adapted KDQoL-SF questionnaire)(max score 130),
13. Quality of life change (at 4 weeks of intervention period and week 8 of study)(mean THERANOVA-500 vs mean REVACLEAR-400)(all subjects) assessed by adapted KDQoL-SF (max score 130),
14. Quality of life change (pre and at 2 weeks of intervention period)(mean THERANOVA-500 vs mean REVACLEAR-400)(all subjects)(assessed by EQ-5D questionnaire)(max score 125),
15. Quality of life change (pre and at 4 weeks of intervention period)(mean THERANOVA-500 vs mean REVACLEAR-400)(all subjects)(assessed by EQ-5D questionnaire)(max score 125),
16. Quality of life change (at 4 weeks of intervention period and week 8 of study)(mean THERANOVA-500 vs mean REVACLEAR-400)(all subjects)(assessed by EQ-5D questionnaire (max score 125),
17. Quality of life change (pre and at 2 weeks of intervention period (mean THERANOVA-500 vs mean REVACLEAR-400)(all subjects)(assessed by rESAS)(max score 100),
18. Quality of life change (pre and at 4 weeks of intervention period (mean THERANOVA-500 vs mean REVACLEAR-400)(all subjects)(assessed by rESAS)(max score 100),
19. Quality of life change (at 4 weeks of intervention period and week 8 of study)(mean THERANOVA-500 vs mean REVACLEAR-400)(all subjects)(assessed by rESAS)(max score 100),
20. Subjects's QoL questionnaire fill preference (adapted KD QoL-SF vs EQ-5D vs rESAS) at study week 8.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years, all genders.
* HD at DrGLDUHC for more than 3 months, 3 times/week schedule, and using REVACLEAR-400.
* Good vascular access (blood flow (Qb) > 300 during entire previous 6 HD sessions, no per-HD alteplase treatments used over the last 2 weeks, routine alteplase-lock allowed)
* Signed informed consent
* Likely to be able to participate for the duration of the clinical evaluation (no trips, no elective procedures, no transfer to another dialysis modality or HD facility, etc).
* Able to fill questionnaires, staff assistance allowed.

Exclusion Criteria:

* HD more than 3 times/week
* HD on other dialyzers than REVACLEAR-400
* Poor vascular access (from staff and Nephrologists' evaluation)
* No consent or unable to answer questionnaires even with staff assistance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2021-06-04 (Estimated)

PRIMARY OUTCOMES:
Post-dialysis recovery time (intervention period) | through 6-week intervention period
  All subjects are asked weekly on their mid-week session how long did it take them to recover from their previous hemodialysis session for the entire duration of the project (10 weeks). Mean post-dialysis recovery time report (in hours) of all subjects on THERANOVA-500 (5 reports/subject) compared to mean of all subjects on REVACLEAR-400 reports during the 6-week intervention period (5 reports/subject) is the primary outcome measure.(intended statistical test: 2-sample t-Test)(re continuous data, n=35/group)

SECONDARY OUTCOMES:
Post-hemodialysis recovery time change (THERANOVA-500 vs REVACLEAR-400) | through 10-week study
  This outcome refers to the mean post-hemodialysis recovery time reports (in hours) during 6-week intervention period (5 reports/subject) minus mean post-hemodialysis recovery time reports of 2-week pre and 2-week post intervention period (5 reports/subject)(all subjects)(intended statistical test: paired t-Test)(re continuous data, n=35/group)
Post-hemodialysis recovery time difference (THERANOVA-500) | through 6-week intervention period
  This outcome refers to the mean difference between blinded and non-blinded THERANOVA-500 treated subjects of post-hemodialysis recovery time (in hours) during the 6-week intervention period (5 reports/subject)(intended statistical test: Wilcoxon Rank Sum Test)(re continuous data, n <= 25/group). This outcome is to assess extent of placebo effect.
Post-hemodialysis recovery time difference (REVACLEAR-400) | through 6-week intervention period
  This outcome refers to the mean difference between blinded and non-blinded REVACLEAR-400 treated subjects of post-hemodialysis recovery time (in hours) during the 6-week intervention period (5 reports/subject)(intended statistical test: Wilcoxon Rank Sum Test)(re continuous data, n <= 25/group). This outcome is to assess extent of placebo effect.
Post-hemodialysis recovery time difference mean gap (THERANOVA-500 vs REVACLEAR-400) | through 6-week intervention period
  This outcome refers to comparison between mean difference of secondary outcome 3 and mean of secondary outcome 4 of post-hemodialysis recovery time (in hours)(intented statistical test: 2-sample t-Test)(re mean of means). This outcome is to assess extent of differential placebo effects between the intervention groups.
Percentage of subjects who report no (zero) recovery time (THERANOVA-500 vs REVACLEAR-400) | through 6-week intervention period
  This outcome refers to the mean difference of percentage of subjects reporting no (zero) recovery time after treatment with THERANOVA-500 compared to mean percentage of subjects reporting no (zero) recovery time after treatment with REVACLEAR-400 during the 6-week intervention period (all subjects)(intended statistical test: 2-sample t-TEST (re continuous data, n = 35/group)
Pre and post 6-week intervention period pre-dialysis levels of beta-2 microglobulin | 6 weeks
  This outcome refers to the mean difference between pre-dialysis levels of beta-2 microglobulin (in nmol/L) (assay: immunoturbidimetry) pre-intervention period compared to post 6-week intervention period between all subjects treated with THERANOVA-500 and all subjects treated with REVACLEAR-400 (intended statistical test: paired t-Test (re continuous data, n = 35/group)
Pre and post 6-week intervention period pre-dialysis levels of procalcitonin | 6 weeks
  This outcome refers to the mean difference between pre-dialysis levels of procalcitonin (in ng/ml) (assay: ELFA (Enzyme-Linked Fluorescent Assay) pre-intervention period compared to post 6-week intervention period between all subjects treated with THERANOVA-500 and all subjects treated with REVACLEAR-400 (intended statistical test: paired t-Test (re continuous data, n = 35/group)
Pre and post 6-week intervention period pre-dialysis levels of free light chains | 6 weeks
  This outcome refers to the mean difference between pre-dialysis levels of free light chains (gamma and lambda) (in mg/L) (assay: immunoturbidimetry) pre-intervention period compared to post 6-week intervention period between all subjects treated with THERANOVA-500 and all subjects treated with REVACLEAR-400 (intended statistical test: paired t-Test (re continuous data, n = 35/group)
Pre and post 6-week intervention period pre-dialysis levels of interleukine-6 | 6 weeks
  This outcome refers to the mean difference between pre-dialysis levels of interleukine-6 (in pg/ml) (assay: ELISA) pre-intervention period compared to post 6-week intervention period between all subjects treated with THERANOVA-500 and all subjects treated with REVACLEAR-400 (intended statistical test: paired t-Test (re continuous data, n = 35/group)
Pre and post 6-week intervention period pre-dialysis levels of C reactive protein | 6 weeks
  This outcome refers to the mean difference between pre-dialysis levels of C reactive protein (in mg/L) (assay: Heterogeneous enzyme immunoassay) pre-intervention period compared to post 6-week intervention period between all subjects treated with THERANOVA-500 and all subjects treated with REVACLEAR-400 (intended statistical test: paired t-Test (re continuous data, n = 35/group)
Quality of life (QoL) change (pre and at 2 weeks of intervention period)(adapted KDQoL-SF) | 2 weeks
  This outcome refers to the mean difference between QoL assessed by adapted KDQoL-SF questionnaire (max score 130, higher better) pre-intervention period compared to post 2-week intervention period between all subjects treated with THERANOVA-500 and all subjects treated with REVACLEAR-400 (intended statistical test: paired t-Test (re continuous data, n = 35/group). This questionnaire is a locally validated adapted version of KDQoL-SF, Version 1.3, Copyright, RAND 1995,1996,1997, available in English and French.
Quality of life (QoL) change (pre and at 4 weeks of intervention period)(adapted KDQoL-SF) | 4 weeks
  This outcome refers to the mean difference between QoL assessed by adapted KDQoL-SF questionnaire (max score 130, higher better) pre-intervention period compared to post 4-week intervention period between all subjects treated with THERANOVA-500 and all subjects treated with REVACLEAR-400 (intended statistical test: paired t-Test (re continuous data, n = 35/group). This questionnaire is a locally validated adapted version of KDQoL-SF, Version 1.3, Copyright, RAND 1995,1996,1997, available in English and French.
Quality of life (QoL) change (at 4 weeks of intervention period and week 8 of study)(adapted KDQoL-SF) | 4 weeks
  This outcome refers to the mean difference between QoL assessed by adapted KDQoL-SF questionnaire (max score 130, higher better) at 4-week intervention period and week 8 of study between all subjects treated with THERANOVA-500 and all subjects treated with REVACLEAR-400 (intended statistical test: paired t-Test (re continuous data, n = 35/group). This questionnaire is a locally validated adapted version of KDQoL-SF, Version 1.3, Copyright, RAND 1995,1996,1997, available in English and French.
Quality of life (QoL) change (pre and at 2 weeks of intervention period)(EQ-5D) | 2 weeks
  This outcome refers to the mean difference between QoL assessed by EQ-5D questionnaire (max score 125, higher better) pre-intervention period compared to post 2-week intervention period between all subjects treated with THERANOVA-500 and all subjects treated with REVACLEAR-400 (intended statistical test: paired t-Test (re continuous data, n = 35/group). This questionnaire is a common validated instrument by EuroQol group available in multiple languages used here in its English and French Canadian versions.
Quality of life (QoL) change (pre and at 4 weeks of intervention period)(EQ-5D) | 4 weeks
  This outcome refers to the mean difference between QoL assessed by EQ-5D questionnaire (max score 125, higher better) pre-intervention period compared to post 4-week intervention period between all subjects treated with THERANOVA-500 and all subjects treated with REVACLEAR-400 (intended statistical test: paired t-Test (re continuous data, n = 35/group). This questionnaire is a common validated instrument by EuroQol group available in multiple languages used here in its English and French Canadian versions.
Quality of life (QoL) change (at 4 weeks of intervention period and week 8 of study)(EQ-5D) | 4 weeks
  This outcome refers to the mean difference between QoL assessed by EQ-5D questionnaire (max score 125, higher better) at 4-week intervention period and week 8 of study between all subjects treated with THERANOVA-500 and all subjects treated with REVACLEAR-400 (intended statistical test: paired t-Test (re continuous data, n = 35/group). This questionnaire is a common validated instrument by EuroQol group available in multiple languages used here in its English and French Canadian versions.
Quality of life (QoL) change (pre and at 2 weeks of intervention period)(rESAS) | 2 weeks
  This outcome refers to the mean difference between QoL assessed by rESAS questionnaire (max score 100, higher better) pre-intervention period compared to post 2-week intervention period between all subjects treated with THERANOVA-500 and all subjects treated with REVACLEAR-400 (intended statistical test: paired t-Test (re continuous data, n = 35/group). This questionnaire is the revised Edmonton Symptom Assessment System instrument available in English and in French.
Quality of life (QoL) change (pre and at 4 weeks of intervention period)(rESAS) | 4 weeks
  This outcome refers to the mean difference between QoL assessed by rESAS questionnaire (max score 100, higher better) pre-intervention period compared to post 4-week intervention period between all subjects treated with THERANOVA-500 and all subjects treated with REVACLEAR-400 (intended statistical test: paired t-Test (re continuous data, n = 35/group). This questionnaire is the revised Edmonton Symptom Assessment System instrument available in English and in French.
Quality of life (QoL) change (at 4 weeks of intervention period and week 8 of study)(rESAS) | 4 weeks
  This outcome refers to the mean difference between QoL assessed by rESAS questionnaire (max score 100, higher better) at 4-week intervention period and week 8 of study between all subjects treated with THERANOVA-500 and all subjects treated with REVACLEAR-400 (intended statistical test: paired t-Test (re continuous data, n = 35/group). This questionnaire is the revised Edmonton Symptom Assessment System instrument available in English and in French.
Subjects's QoL questionnaire fill preference | at week 10 of study
  At the end of the study (week 10) all subjects will be asked which QoL questionnaire (between the adapted KDQoL-SF, EQ-5D and rESAS) they prefer to fill for future routine use in the hemodialysis unit.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Dorval, MD,MPH,MBA, Principal Investigator — Dr Georges-L.-Dumont University Hospital Centre
Locations (1):
- Dr Georges-L.-Dumont University Hospital Centre, Moncton, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: No
This is no plan to share individual participant data as this was not approved by local ethic review board.